CLINICAL TRIAL: NCT03703245
Title: A Post-hoc Pooled Analysis of GSK CH Clinical Data Investigating the Efficacy of a Dentifrice Containing 67% w/w Sodium Bicarbonate on Gingivitis and Plaque Accumulation
Brief Title: Pooled Analysis of Clinical Data From Six GSK Studies to Investigate the Efficacy of a Dentifrice Containing 67% Weight by Weight (w/w) Sodium Bicarbonate on Gingivitis and Plaque Accumulation
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 209509
Record Dates: First submitted 2018-09-14; First posted 2018-10-11 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Gingivitis; Dental Plaque
Keywords: Plaque Accumulation
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — Sodium Bicarbonate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Dentifrice: Participants were advised to brush their teeth twice daily with a full strip of experimental dentifrice containing 67% w/w sodium bicarbonate in 3 studies and additionally 62% w/w sodium bicarbonate in 3 studies covering the entire head of the toothbrush for 1 minute.
  Interventions: Other: Sodium bicarbonate
- Control Dentifrice: Participants were advised to brush their teeth with control dentifrice containing 0% w/w sodium bicarbonate covering the entire head of the toothbrush for 1 minute.
  Interventions: Other: Control Dentifrice

INTERVENTIONS:
Other: Sodium bicarbonate — Experimental dentifrice containing 67% w/w sodium bicarbonate in 3 studies and additionally 62% w/w sodium bicarbonate in 3 studies.
  Groups: Experimental Dentifrice
Other: Control Dentifrice — Negative control dentifrice containing 0% w/w sodium bicarbonate
  Groups: Control Dentifrice

SUMMARY:
The aim of this analysis was to pool data from 6 GSK studies with similar clinical design to investigate the overall efficacy of a test dentifrice containing 67% w/w sodium bicarbonate in the treatment of gingivitis and plaque accumulation after 6, 12 and 24 weeks of twice-daily brushing at home relative to a negative control dentifrice.

The pooled analysis was planned and conducted after completion of all six independent studies.

DETAILED DESCRIPTION:
This pooled analysis was performed on data collated from six GSK studies that provide efficacy data supporting the twice-daily use of a dentifrice containing 67% w/w sodium bicarbonate in the management of pre-existing gingivitis, and plaque accumulation. Six studies that were chosen for inclusion in the pooled analysis were single-center, examiner-blind, 2 to 3 treatments, parallel group, stratified and randomized clinical study. In all studies, participants entered the screening period during which eligibility for the study was determined. The participants included male and non-pregnant, non-lactating female subjects at least 18 years of age with pre-existing gingivitis as determined by an appropriately qualified clinical examiner. Participants meeting the inclusion criteria entered an acclimatization period in order to minimize any potential placebo response. Participants were randomized into treatments, parallel group, stratified and randomized clinical studies twice daily at home for 6, 12 and 24 weeks and participants returned to the site. Participants underwent a full OST examination and the recording of any Adverse Events (AEs). Participants then underwent Modified Gingival Index (MGI), Bleeding Index (BI), Gingival Severity Index (GSI) followed by dental plaque assessments.

ELIGIBILITY:
Inclusion Criteria:

* Clinical studies conducted by GSK CH, including access to study protocols, study reports, and access to individual information sources/ study data.
* Study design and subject inclusion criteria in agreement with guidelines to assess gingivitis efficacy such as inclusion of a pre-treatment full-mouth prophylaxis, Subject eligibility (>20 bleeding sites and mild-moderate gingivitis at Screening);Comparable indices of gingivitis and plaque accumulation; a treatment for a 67% w/w sodium bicarbonate dentifrice; Repeat brushing for at least a period of 4 weeks or 4-6 weeks.

Exclusion Criteria: Not Applicable

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retrospective pooled studies include healthy male and non-pregnant, non-lactating female subjects at least 18 years of age, with pre-existing gingivitis as determined by an appropriately qualified clinical examiner
Sampling Method: Probability Sample
Enrollment: 1601 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Mean number of Bleeding Sites over 24 weeks | Over 24 weeks
  Number of gingival bleeding sites were measured as BI via a single examiner using a color coded periodontal probe. The probe was gently inserted approximately 1 millimeter (mm) into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. The BI scoring system used to measure bleeding sites is as follows: 0= No bleeding after 30 seconds; 1= Bleeding upon probing after 30 seconds; 2= Immediate bleeding observed. A bleeding site was considered as a BI score of 1 or 2. This measure will be analyzed and summarized over all sites and at the tooth site level.

SECONDARY OUTCOMES:
Mean Bleeding Index (BI) over 24 weeks | Over 24 weeks
  The BI was performed by a single examiner using a color coded periodontal probe. The probe was inserted approximately 1 mm into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. The BI scoring system to be used is as follows: 0= No bleeding after 30 seconds; 1= Bleeding upon probing after 30 seconds; 2= Immediate bleeding observed. This measure will be analyzed and summarized over all sites and at the tooth site level.
Mean Modified Gingival Index (MGI) over 24 weeks | Over 24 weeks
  The MGI was assessed on facial and lingual surfaces at two sites on each tooth (papillae and margin).The scoring of MGI was performed by a single examiner. The MGI scoring system is as follows:0=absence of inflammation;1=mild inflammation; slight change in color, little change in color;little change in texture of any portion of the marginal or papillary gingival unit;2=mild inflammation; criteria as above but involving the entire marginal or papillar gingival units;3=moderate inflammation; glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit;4=severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration.This measure will be analyzed and summarized over all sites and at the tooth site level.
Mean Turesky modification of the Quigley Hein plaque index (TPI) over 24 weeks | Over 24 weeks
  The dental examiner used the TPI to assess plaque on all gradable teeth. The plaque was first disclosed using a dye solution. Participants then rinsed with disclosing solution according to instructions. They had expectorated and rinsed with 10 mL of water for 10 seconds and expectorated again. Plaque was assessed with each tooth being divided into 6 areas including the mesiofacial, facial, distofacial, mesiolingual, lingual and distolingual surfaces. Disclosed plaque was scored as follows: 0= No plaque; 1= Slight flecks of plaque at the cervical margin of the tooth; 2= A thin continuous band of plaque (1 mm or smaller) at the cervical margin of the tooth; 3= A band of plaque wider than 1 mm but covering less than 1/3 of the crown of the tooth; 4= Plaque covering at least 1/3 but less tan 2/3 of the crown of the tooth; 5= Plaque covering 2/3 or more of the crown of the tooth.This measure will be analyzed and summarized over all sites and at the tooth site level.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Weybridge, Surrey, United Kingdom